CLINICAL TRIAL: NCT03715764
Title: Physical Therapist as Primary Assessor for Patients With Knee Pain in Primary Health Care. A Randomized Controlled Study
Brief Title: Physical Therapist as Primary Assessor for Patients With Knee Pain in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115841rct
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2018-10

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Physical Therapist; Primary assessor; Primary care
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy assessment (Other): Patients allocated to the intervention group will be assigned to an assessment and evaluation by a physical therapist. If they are diagnosed with knee osteoarthritis they will get an offer to participate in a patient education program and physical training with an individualized exercise program made by a physical therapist. Patients will be offered individual treatment if they decline to participate in the education program, or if they have another diagnosis than osteoarthritis. Anytime after the first assessment by the physical therapist, the patient will be able to contact a physician if they want to.
  Interventions: Other: Physical therapy assessment
- Physician assessment (Other): Allocation to the control group will involve an assessment and evaluation made by a physician. Further measures will then be determined by attending physician and the procedures that might get included are drug prescriptions, referral to x-ray examination, referral to a physical therapist or another health care provider. Anytime after the first assessment by the physician, the patient will be able to contact a physical therapist if they want to, even though if they have not been referred by the physician.
  Interventions: Other: Physician assessment

INTERVENTIONS:
Other: Physical therapy assessment — Primary assessment, diagnose and treatment by a physical therapist for patients with knee pain in primary care.
  Arms: Physical therapy assessment
Other: Physician assessment — Primary assessment, diagnose and treatment by a physician for patients with knee pain in primary care.
  Arms: Physician assessment

SUMMARY:
In order to manage the future increase in osteoarthritis consultation, patients with osteoarthritis could be assessed by a physical therapist first, so that other patients with more severe conditions could get faster access to a primary care physician. In Swedish primary care, physicians and physical therapists are primary assessors for patients with suspected knee osteoarthritis. However, it is unclear if there are any differences between these managements in improving health-related quality of life (HrQoL), pain, physical function and self-efficacy.

There are a limited amount of studies about the impact on HrQoL, pain intensity, self-efficacy and physical performance in patients with knee pain being assessed and evaluated by a physical therapist as a primary assessor.

The overall purpose of this study is to evaluate the effects on self-rated HrQoL, pain intensity, self-efficacy and physical performance with either a physical therapist or a physician as primary assessor for patients with knee pain within primary health care.

Problem statements

Which effect does a clinical pathway with a physical therapist as primary assessor for patients with knee pain…

1. … have on self-rated HrQoL compared with a physician as primary assessor?
2. … have on self-rated pain intensity compared with a physician as primary assessor?
3. … have on physical performance compared with a physician as primary assessor?
4. … have on self-efficacy compared with a physician as primary assessor?

It is expected that this study will show the effects of two different primary assessors for patients with knee pain consulting primary health care. The results could clarify which profession that is most appropriate to be the primary assessor for patients with knee pain in primary health care.

DETAILED DESCRIPTION:
Patient Recruitment Recruiters: Primary care centers.

Screening procedure: Nurses at the primary care centers will get information about the study and the screening protocol from the data collector and project leader. There will be contact persons at each recruiting unit that will be responsible for the protocols and to contact the data collector when a patient fulfills all the criteria for participation. The project leader will have regular contact with the contact persons at the recruiting units. All screening protocols will be sent to the data collector. All participants will get orally and written information about the study from the data collector, and patients will provide written informed consent.

Randomization: Using a computer-generated list of random numbers, participants will be randomly assigned to being assessed, diagnosed and treated either by a physiotherapist or a physician first. A project coordinator is included among the health care providers in the study, but will not be involved in the screening procedure nor the data collection. The project coordinator will manage the sequence generation, allocation concealment, enrolment and assignments of participants and keep the concealed randomization scheme and sequentially numbered, sealed envelopes in a locked cupboard (in the same building where the enrolment will be), only available for the project coordinator. The project coordinator reveals the allocation to the participant shortly after the baseline measurement and to the health care providers.

Participants and health care providers in both groups will be aware of the allocated group, whereas data collector, data analyst and statistician will be kept blinded of allocation until completion of all outcome assessments.

The blinded data collector and analyst (is a physical therapist) whom is not involved in assessing diagnosing and treating patients with knee osteoarthritis while the study is conducted.

Data Collection: Measurements will be collected at baseline (before randomization), at 3- , 6- , and at 12 months follow up.

Data management: All data will be coded and managed according to the Data Protection Act (1998:204), which means that all data will be confidential and no unauthorized will have access to the patient registry. The results will be presented at group level, therefore, no individual information can be identified. Data will be saved for at least 10 years to enable audit.

Sample size: To detect a minimal clinical improvement in health related quality of life of 0.121(SD 0.2) on the EQ5D-index, with a two-sided 5% significance level and a power of 80%, a sample size of 50 patients per group will be necessary, given an anticipated dropout rate of 14%.

Statistical analysis: Data will be analyzed descriptively and presented as numbers and percent, mean and standard deviation or median and 25th to 75th percentiles. The primary outcome will be mean change in HrQoL (EQ5D-index and EQ5D-scale) and secondary outcomes will include mean change in pain intensity (VAS), physical performance (30CST) and self-efficacy (ASES-S). The changes in scores for the outcomes will be constructed by calculating raw differences between baseline and the follow ups. For group comparison the Χ2-test will be used for nominal data and Fischer's exact test for small numbers, parametric student t-test for continuous variables and Mann-Whitney's test for ordinal data and at skewed distributions. Statistical analysis will be made in SPSS Windows and the analysis will be applied with intention-to-treat (ITT). The level of significance will be p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age >38 years old
* Knee pain most of the days the last month
* Crepitus on active motion
* Morning stiffness, duration less than 30 minutes
* The patient has to understand the Swedish language to follow test instructions and to complete the self-administered questionnaires.

Exclusion Criteria:

* Already been assessed/diagnosed by a healthcare provider for current knee pain.
* knee pain due to a traumatic cause
* other rheumatic or systemic diseases
* severe somatic or mental disease
* pregnancy.

Min Age: 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Nordeman, RPT, PhD, Principal Investigator — Research & Development Centre Södra Älvsborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turkiewicz A, Petersson IF, Bjork J, Hawker G, Dahlberg LE, Lohmander LS, Englund M. Current and future impact of osteoarthritis on health care: a population-based study with projections to year 2032. Osteoarthritis Cartilage. 2014 Nov;22(11):1826-32. doi: 10.1016/j.joca.2014.07.015. Epub 2014 Jul 30. PMID 25084132
- [Background] Walters SJ, Brazier JE. Comparison of the minimally important difference for two health state utility measures: EQ-5D and SF-6D. Qual Life Res. 2005 Aug;14(6):1523-32. doi: 10.1007/s11136-004-7713-0. PMID 16110932
- [Background] Brazier JE, Harper R, Munro J, Walters SJ, Snaith ML. Generic and condition-specific outcome measures for people with osteoarthritis of the knee. Rheumatology (Oxford). 1999 Sep;38(9):870-7. doi: 10.1093/rheumatology/38.9.870. PMID 10515649
- [Background] Fransen M, Edmonds J. Reliability and validity of the EuroQol in patients with osteoarthritis of the knee. Rheumatology (Oxford). 1999 Sep;38(9):807-13. doi: 10.1093/rheumatology/38.9.807. PMID 10515639
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Gill SD, de Morton NA, Mc Burney H. An investigation of the validity of six measures of physical function in people awaiting joint replacement surgery of the hip or knee. Clin Rehabil. 2012 Oct;26(10):945-51. doi: 10.1177/0269215511434993. Epub 2012 Feb 9. PMID 22324057
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Derived] Ho CM, Thorstensson CA, Nordeman L. Physiotherapist as primary assessor for patients with suspected knee osteoarthritis in primary care-a randomised controlled pragmatic study. BMC Musculoskelet Disord. 2019 Jul 13;20(1):329. doi: 10.1186/s12891-019-2690-1. PMID 31301739

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assessed for eligibility (n=363)
  Excluded (n=294)
  * Not meeting inclusion criteria (n=185)
  * Declined to participate (n=15)
  * Excluded due to exclusion criteria (n=94)
Period: Baseline (Randomized (n=69)
Arm/Group | Physical Therapy Assessment | Physician Assessment
Started | 35 | 34
Completed | 33 | 31
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3
Period: 3 Month Follow-up
Arm/Group | Physical Therapy Assessment | Physician Assessment
Started | 33 | 31
Completed | 30 | 28
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Period: 6 Month Follow-up
Arm/Group | Physical Therapy Assessment | Physician Assessment
Started | 30 | 28
Completed | 27 | 28
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0
Period: 12 Month Follow-up
Arm/Group | Physical Therapy Assessment | Physician Assessment
Started | 27 | 28
Completed | 21 | 23
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Surgery | 2 | 0
Not completed — Wrong address | 1 | 0
Not completed — No symptoms | 1 | 0
Not completed — Changed primary care centre | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Therapy Assessment | Physician Assessment | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.6) | 59 (11.5) | 60 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 14 | 11 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Level of education [Count of Participants; unit: Participants]
  Primary school | 8 | 4 | 12
  Secondary school | 15 | 20 | 35
  Tertiary school | 12 | 10 | 22
Current Employment [Count of Participants; unit: Participants]
  Employed/working | 19 | 18 | 37
  Unemployed | 0 | 1 | 1
  Retired/early retirement | 15 | 13 | 28
  Sick leave | 1 | 2 | 3
Pain duration (months) [Mean (Standard Deviation); unit: months] | 14 (22) | 10 (16) | 12 (19)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30 (4.4) | 29 (6.7) | 29 (5.6)
Health-related quality of life (EQ5D-index) [Mean (Standard Deviation); unit: units on a scale] — The questionnaire contain five dimensions and results is an index ranging from -0,549 to 1 using the UK tariffs. An index of 1 indicate full health.
  units on a scale | 0.73 (0.121) | 0.62 (0.222) | 0.67 (0.185)
Health-related quality of life (EQ5D-VAS) [Mean (Standard Deviation); unit: units on a scale] — The EQ5D-VAS is a visual analogue scale ranging from 0 to 100, where 0 is worst imaginable health state and 100 is best imaginable health state.
  units on a scale | 73 (17.5) | 68 (21.1) | 70 (19.5)
Pain intensity (VAS 0-100) [Mean (Standard Deviation); unit: units on a scale.] — 0=no pain, 100=worst imaginable pain
  units on a scale. | 45 (15.9) | 52 (16.4) | 49 (16.5)
Physical function (30 CST) [Mean (Standard Deviation); unit: Chair stands] — Physical performance were measured with 30 seconds chair stand test (30CST). Number of chair stands were counted.
  Chair stands | 12 (4.6) | 11 (3.3) | 12 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Health Related Quality of Life (HrQoL) at 12 Months - EQ5D-index
Description: A Swedish version of Euroqol-5 dimensions-3 levels (EQ5D-3L) will be used to assess perceived self-rated health-related quality of life. The questionnaire contain five dimensions and results in an index ranging from -0,549 to 1 using the UK tariffs. An index of 1 indicate full health.
Time Frame: 12 months
Population: Mixed effect model analyses were used to compare the repeated measures of HrQoL between groups. Presenting the estimated marginal means for the final model (adjusted for confounders) at the 12 month follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Physical Therapy Assessment | Physician Assessment
Number analyzed (Participants) | 35 | 34
score on a scale | 0.804 (0.025) | 0.825 (0.024)
Statistical Analysis 1: Comparison: Physical Therapy Assessment vs Physician Assessment; Test type: Superiority; p = 0.87, Mixed Models Analysis — Results for the final model, variable GROUP, adjusted for confounders
Statistical Analysis 2: Comparison: Physical Therapy Assessment vs Physician Assessment; Test type: Superiority; p < 0.001, Mixed Models Analysis — Results for the final model for the variable TIME, adjusted for confounders
Statistical Analysis 3: Comparison: Physical Therapy Assessment vs Physician Assessment; Test type: Superiority; p = 0.18, Mixed Models Analysis — Results for the final model, variable Group x Time (Statistical interaction of group and time), adjusted for confounders

2. Primary Outcome: Change From Health Related Quality of Life (HrQoL) at 12 Months - EQ5D-VAS
Description: A Swedish version of Euroqol-5 dimensions-3 levels (EQ5D-3L) will be used to assess perceived self-rated health-related quality of life. The EQ5D-VAS is a visual analogue scale ranging from 0 to 100, where 0 is worst imaginable health state and 100 is best imaginable health state.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Physical Therapy Assessment | Physician Assessment
Number analyzed (Participants) | 35 | 34
score on a scale | 81 (2.55) | 77 (2.49)
Statistical Analysis 1: Comparison: Physical Therapy Assessment vs Physician Assessment; Test type: Superiority; p = 0.56, Mixed Models Analysis — Results for the final model, variable GROUP, adjusted for confounders
Statistical Analysis 2: Comparison: Physical Therapy Assessment vs Physician Assessment; Test type: Superiority; p = 0.0049, Mixed Models Analysis — Results for the final model, variable TIME, adjusted for confounders
Statistical Analysis 3: Comparison: Physical Therapy Assessment vs Physician Assessment; Test type: Superiority; p = 0.49, Mixed Models Analysis — Results for the final model, adjusted for confounders, for the variable Group x Time (Statistical interaction of group and time)

3. Secondary Outcome: Change From Pain Intensity at 12 Months
Description: The mean pain intensity (over the past month) will be measured by a visual analogue scale (VAS) ranged from 0 which will correspond no pain and 100 the worst imagined pain.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Therapy Assessment | Physician Assessment
Number analyzed (Participants) | 19 | 17
units on a scale | 21.79 (18.59) | 23.29 (18.87)
Statistical Analysis 1: Comparison: Physical Therapy Assessment vs Physician Assessment; Test type: Superiority — Used as a confounder in the mixed effect model analysis for primary outcome. All participants enrolled in the study were included in the 12 months analysis; p < 0.2, Mixed Models Analysis — Confounding variables with p-values < 0.2 were carried forward to the final model

4. Secondary Outcome: Change From Physical Function at 12 Months
Description: Physical performance will be measured with 30 seconds chair stand test (30CST). Number of chair stands will be counted.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: stands
Arm/Group | Physical Therapy Assessment | Physician Assessment
Number analyzed (Participants) | 19 | 22
stands | 15 (4.9) | 15 (5.8)
Statistical Analysis 1: Comparison: Physical Therapy Assessment vs Physician Assessment; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.2, Mixed Models Analysis — Confounding variables with p-values < 0.2 were carried forward to the final model

5. Secondary Outcome: Change From Self-efficacy at 12 Months
Description: Self-efficacy will be assessed with Arthritis Self-Efficacy Scale-Swedish version (ASES-S). Each question range from 10-100, where 10 is very insecure and 100 is very confident. The questionnaire consists three subscales in how patients are experiencing their 1) pain, 2) physical function, 3) other symptoms. Each subscale results in a mean score ranging from 10 to 100 where 10 means very insecure and 100 means very confident.
  The results of this outcome measure has not been analysed for publication. This outcome measure were excluded in the first manuscript when submitted to scientific journal and will probably be reported in a second manuscript. Anticipated reporting date is December 2024.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Physical Therapy Assessment | Physician Assessment
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

LIMITATIONS AND CAVEATS:
* Due to low participant inflow, the recruting was ended before reaching the required sample size of 100 patients.
* Under powered study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT03715764/Prot_SAP_000.pdf